CLINICAL TRIAL: NCT05559229
Title: Poorly Differentiated Adenocarcinoma With Signet Ring Cells of the Gallbladder Producing a High Level of Alpha-fetoprotein: a Case Report
Status: Completed | Type: Observational
Sponsor: junya mita (Other)
Responsible Party: Sponsor-Investigator, junya mita, principal investigator, Oita Red Cross Hospital
Organization: Oita Red Cross Hospital (Other)
Other Study IDs: oitaRCH
Record Dates: First submitted 2022-09-19; First posted 2022-09-29 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Gallbladder Cancer
MeSH Terms: conditions — Gallbladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: laparoscopic whole-layer cholecystectomy — laparoscopic whole-layer cholecystectomy.

SUMMARY:
Alpha-fetoprotein (AFP) can become elevated in hepatocellular carcinoma (HCC), yolk sac tumors and other malignant tumors of various organs. Herein, the investigator present a case of AFP-producing gallbladder carcinoma with signet ring cells successfully treated with laparoscopic whole-layer cholecystectomy.

ELIGIBILITY:
The study eligibility criteria for patient were as follows: AFP-producing gallbladder carcinoma (cT2aN0M0, cStage IIa, UICC 8th) or gallbladder metastasis from HCC.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: a case of AFP-producing gallbladder carcinoma with signet ring cells
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2022-06-25 (Actual); Study Completion 2022-09-18 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of measuring value of AFP for patients with gallbladder cancer. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- oita Red Cross hospital, Ōita, Oita Prefecture, Japan

IPD SHARING:
Plan to Share IPD: No